CLINICAL TRIAL: NCT06983041
Title: Open-label, Uncontrolled Clinical Research Study of a Vaginal Cooling Device for the Treatment of Vulvovaginal Candidiasis (VVC)
Brief Title: Clinical Study of a Vaginal Cooling Device for the Treatment of Vulvovaginal Candidiasis (VVC)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Coologics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00079644
Record Dates: First submitted 2025-05-02; First posted 2025-05-21 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Vulvovaginal Candidiasis (VVC); Yeast Vaginitis
Keywords: yeast infection
MeSH Terms: conditions — Candidiasis, Vulvovaginal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- uncomplicated vulvovaginal candidiasis (Other): Twice daily use of vaginal cooling device for 30 minutes a time for three days (i.e., 3 hours total) in female subjects with VVC age 22-49 (inclusive).
  Interventions: Device: vaginal cooling device

INTERVENTIONS:
Device: vaginal cooling device — medical grade polymer capsule filled with inert fluid (15 cc's)

SUMMARY:
The objective of this study is to determine clinical cure rate and safety of a proprietary Vaginal Cooling Device (VCD) in women with VCC. In addition, the safety, mycological cure rates, the speed and efficacy of symptom resolution, vaginal hyphae and polymorphonuclear (PMN) scores, and Quality-of-Life (QoL) parameters will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Site investigators will evaluate the eligibility of women presenting with symptoms consistent with VVC based on the inclusion criteria.

  1. Women between 22-49 years of age and not more than one year since last menses, with the suspected diagnosis of uncomplicated VVC.
  2. Able to read and understand English.
  3. Able to provide written informed consent and to understand and agree to all study procedures required.
  4. Has a smart phone and has the ability to access and use the ValidCare app.
  5. Documented Papanicolaou (Pap) test at baseline or during the previous 12 months reported as either "negative for intraepithelial lesion or malignancy" or "ASCUS-atypical squamous cells of undetermined significance" and negative for high-risk HPV types or negative colposcopy plus/minus biopsies were performed for high-risk HPV types.
  6. Clinical diagnosis of symptomatic VVC confirmed by positive KOH wet mount and yeast culture at baseline.
  7. Presence of at least one vulvovaginal sign (vulvovaginal erythema, edema, or excoriation) of VVC.
  8. Presence of at least one vulvovaginal symptom (itching, pain or burning, irritation)
  9. Willing and able to avoid vaginal (or any) sexual activity during the study period.
  10. Menstrual products such as tampons, pads, and menstrual cups may be used during the study period including before and after device use.

Exclusion Criteria:

* 1. Site investigators will evaluate the eligibility of women presenting with symptoms consistent with VVC based on the exclusion criteria.

  2. Subject does not have a smart phone. 3. Subject does not have the ability to access and use the Validcare app. 4. Subjects who were treated for VVC within the past 14 days. 5. Use of systemic, topical (applied to the vulva) or vaginal antibiotics, anti-fungal or anti-trichomonas drugs within 14 days.

  6. Use of any systemic corticosteroid, immunosuppressive, or immune-stimulating drug within 3 months.

  7. History of douching within the previous 7 days. 8. Urinary tract infection. 9. Unable or unwillingness to use tampons in the past. 10. Unable to maintain study protocol including but not limited to the avoidance of sexual activity during the 28 days or time interval up to the assessment of the primary endpoint. This is needed to avoid reinfection, worsening of symptoms or new pathogen infection, while assessing the efficacy of the subject device in treating the primary infection.

  11. Use of anticoagulation therapy (e.g., warfarin, heparin). 12. Diabetes mellitus. 13. History of vulvodynia, vestibulitis, vaginismus, radiation-induced vaginitis, or postmenopausal atrophy.

  14. Immune compromised states such as HIV/AIDS or transplant subjects. 15. Subjects with other infectious causes of vulvovaginitis or with mixed infections diagnosed at baseline. (Note: if any trichomonad trophozoites are seen on wet smear on the initial visit, the subject is to be excluded from the study.) 16. Symptomatic vulvar or vaginal condyloma or presence of another vaginal or vulvar condition that would confound the interpretation of clinical response.

  17. Pregnancy. 18. Presence of trichomonad trophozoites on wet smear at the initial visit. 19. Any condition which, in the opinion of the investigator, should preclude participation in the study. If so, the investigator will collect information on the subjects who are determined to have a condition that precludes participation in the study and the reasons for their exclusion documented within the DDCS to ensure there is no bias introduced.

Ages: 22 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 55 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of clinical cures at 7 days | 7 days (+/-2)
  VSS of 0-1(based on severity of infection), KOH negative for Hyphae

SECONDARY OUTCOMES:
Clinical Cure | 28 days (+/-2)
  VSS of 0-1(based on severity of infection), KOH negative for Hyphae

OTHER OUTCOMES:
Mycological Cure | 7 days (+/-2)
  Negative fungal culture for offending species
Mycological Cure | 28 days (+/- 2)
  Negative fungal culture for offending species
Polymorphonuclear Neutrophils (PMN) | 7 days (+/-2)
  Quantification of PMNs
Polymorphonuclear Neutrophils (PMN) | 28 days (+/- 2)
  Quantification of PMNs
Hyphae Scores | 7 days (+/-2)
  Quantification of Hyphae levels
Hyphae Scores | 28 days (+/- 2)
  Quantification of Hyphae levels

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Symphony Clinical Research, Jacksonville, Florida
  - Nova Clinical Research, Miami, Florida
  - Pivotal Clinical Research & Associates, Smyrna, Georgia
  - Renew Health Clinical Research, Snellville, Georgia
  - Leavitt Clinical Research, Idaho Falls, Idaho
  - Next Innovative Clinical Research, Chicago, Illinois
  - Unified Women's Clinical Research-Raleigh, Raleigh, North Carolina
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - Aviati Health, Memphis, Tennessee
  - Vilo Research Group, Inc., Houston, Texas

IPD SHARING:
Plan to Share IPD: No